CLINICAL TRIAL: NCT05212077
Title: Effect of Advanced Care at Home vs. Traditional Brick-and-Mortar Hospital Care in Acutely Ill Adults: A Randomized Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Xiaoxi Yao, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-005335
Record Dates: First submitted 2022-01-26; First posted 2022-01-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: The Trial Will Compare Two Care Delivery Models That Are Currently Being Used in Routine Practice Settings for Acute Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Care at Home (ACH) (Experimental): Patients will receive inpatient hospitalization at home.
  Interventions: Other: Advanced Care at Home (ACH)
- Traditional Inpatient (Brick-and-Mortar) Hospital Care (Active Comparator): Patients will receive inpatient hospitalization at the hospital.
  Interventions: Other: Traditional Brick-and-Mortar Hospitalization

INTERVENTIONS:
Other: Advanced Care at Home (ACH) — Inpatient hospitalization offered in the home setting.
  Arms: Advanced Care at Home (ACH)
Other: Traditional Brick-and-Mortar Hospitalization — Inpatient hospitalization offered in the hospital setting.
  Arms: Traditional Inpatient (Brick-and-Mortar) Hospital Care

SUMMARY:
The purpose of this study is to compare two care delivery models that are currently being implemented in routine practice settings. The findings from this study will inform future clinical decision making, such as which patients might be more suited for which care delivery model.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years of age and older.
* Present to one of the participating hospitals.
* Have a chief complaint of one of the target diagnoses.
* Are within a certain geographical area (based on zip codes).
* Have a health insurance plan that covers ACH services.
* Have the capacity to consent or could assent with the consent of a health care proxy who is physically present.

Exclusion Criteria:

* The patient is not suitable for ACH or inpatient hospital care based on:

  * being a nursing home patient;
  * on or requiring dialysis;
  * positive for COVID-19;
  * having discharge order;
  * requiring intensive care unit (ICU) level of care;
  * history of drug abuse.
* Patients will also need to meet the clinical stability criteria.
* Do not have the capacity to consent or assent with the assistance of a health care proxy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a composite outcome of all-cause mortality | 30 days post-discharge
  The rate of death
30-day readmission. | 30 days post-discharge
  readmission between discharge from ACH/traditional inpatient hospital care and 30 days post-discharge.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Mayo Clinic Health System, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao X, Paulson M, Maniaci MJ, Dunn AN, Nelson CR, Behnken EM, Hart MS, Sangaralingham LR, Inselman SA, Lampman MA, Dunlay SM, Dowdy SC, Habermann EB. Effect of hospital-at-home vs. traditional brick-and-mortar hospital care in acutely ill adults: study protocol for a pragmatic randomized controlled trial. Trials. 2022 Jun 16;23(1):503. doi: 10.1186/s13063-022-06430-6. PMID 35710450